CLINICAL TRIAL: NCT05650242
Title: An Non-randomized Open-label, Multicenter Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics, Preliminary Efficacy of BA1106 in Participants With Advanced Solid Tumors
Brief Title: A Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BA1106 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Boan Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA1106/CT-CHN-101
Record Dates: First submitted 2022-11-18; First posted 2022-12-14 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumors
Keywords: BA1106; First in human study; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BA1106 (Experimental): Part A (Dose-Escalation): Mixed solid tumors participants will receive ascending doses of BA1106. BA1106 will be administered by intravenous (IV) infusion. The observation period of Dose Limiting toxicity (DLT) is 28 days, then the participants will receive BA1106 every three weeks (Q3W) until confirmed progression, death, unaccepted toxicity, initiation of other antitumor therapies, or any other conditions requiring treatment discontinuation, and the maximum duration of administration was no more than 2 years.
  Part B (Dose-Expansion): Participants of selected tumors will receive a fixed dose of BA1106 that selected according to the results of Part A once every 3 weeks (Q3W) or once every 2 weeks (Q2W), until confirmed progression, death, unaccepted toxicity, initiation of other antitumor therapies, or any other conditions requiring treatment discontinuation, and the maximum duration of administration was no more than 2 years.
  Interventions: Drug: BA1106

INTERVENTIONS:
Drug: BA1106 — In part A, after the observation period of DLT (28 days), intravenous (IV) once every 3 weeks (Q3W).
  In Part B, intravenous (IV) once every 3 weeks (Q3W) or once every 2 weeks (Q2W).

SUMMARY:
This is an open label Phase 1, First in Human trial designed to evaluate the safety, tolerability pharmacokinetics, preliminary efficacy of BA1106 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
BA1106 is a human anti-CD25 monoclonal antibody. There are two parts in the study. Part A is dose escalation study, and Part B is dose expansion study. Part A will be conducted using BOIN dose escalation method at the dosing regimen of once every 3 weeks. In Part B, 1~2 dose levels, dosing regimens (i.e. once every 2 weeks or once every 3 weeks), and 1~4 selected indications will be chosen to further evaluate the safety and efficacy of BA1106.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the study protocol;
2. Subject with histologically or cytologically confirmed advanced and/or metastatic solid tumors who have progressed on all standard therapies, are intolerant to Standard-Of-Care (SOC), and/or are non-amenable to SOC;
3. At least one evaluable lesion in Part A and at least one measurable lesion in Part B according to RECIST v1.1;
4. Able to provide the most recent archival tumor tissue samples (negotiable);
5. Life expectancy >=12 weeks;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. Adequate major organ function;
8. Women of Childbearing Potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods;
9. Men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods and refrain from donating sperm.

Exclusion Criteria:

1. Participants with active central nervous system (CNS) metastases causing clinical symptoms or metastases that require therapeutic intervention;
2. Participants with any infection requiring intravenous therapy, or any other uncontrolled active infection, within 2 weeks prior to informed consent;
3. Participants with symptomatic radiation pneumonia, radiation esophagitis, radiation colitis; extensive interstitial lung disease of both lungs, chronic obstructive pulmonary disease requiring bronchodilators or regular hormonal therapy; unhealed peptic ulcers, cirrhosis and related complications, chronic enteritis, necrotizing enteritis, gastrointestinal obstruction (except those who are relieved with treatment and have no safety risk as assessed by the investigator), gastrointestinal bleeding tendency or high risk of perforation, pancreatitis requiring treatment; arteriovenous thrombotic disease; chronic nephritis and nephrotic syndrome, within 8 weeks prior to C1D1;
4. Participants with active autoimmune disease or the risk of recurrence;
5. Participants with major cardiocerebral vascular disease;
6. Participants with body cavity effusion requiring local treatment or determined as poorly controlled by the investigator;
7. History of Stevens-Johnson syndrome, toxic epidermal necrolysis, or DIHS (drug-induced hypersensitivity syndrome);
8. Participants with diseases affecting intravenous injection and venous blood collection;
9. Prior use of any anti-cancer therapy (including chemotherapy, radiotherapy, targeted therapy, immunotherapy, traditional Chinese medicine, etc.) within 4 weeks, or non-antitumor traditional Chinese medicine within 2 weeks, prior to C1D1;
10. Prior use of drugs targeting IL-2 receptors;
11. History of being receipt of any organ transplantation or allogeneic stem-cell transplantation;
12. Risk of gastrointestinal ulcers or bleeding as assessed by the investigator;
13. Prior treatment with systemic immunosuppression excluding nasal/inhaled corticosteroids or physiological dosed systemic corticosteroids, within 2 weeks prior to C1D1;
14. Prior treatment with cytokine, blood transfusion, or blood products within 4 weeks prior to C1D1;
15. Participants with major surgical procedure or significant traumatic injury, within 4 weeks prior to C1D1; or with wound healing complications before enrolment;
16. Vaccination with live vaccines within 4 weeks prior to informed consent;
17. Known hypersensitivity to any of the components of BA1106;
18. Participants with grade 2 or higher toxicities from any previous therapies [except for cases of alopecia and peripheral sensory neuropathy (both grade 2), which are allowed];
19. Positive for Hepatitis B and C, or positive HIV test at screening;
20. History of drug abuse, drug addiction, or alcoholism;
21. Pregnancy, lactation, or breastfeeding;
22. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) (according to NCI CTCAE 5.0). | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment, up to 2 years.

SECONDARY OUTCOMES:
Area under the curve (AUC) of BA1106 | up to cycle 6nd (cycle 1st is 28 days, the other cycles are 21 days)
Half-life (t1/2) of BA1106 | up to cycle 6nd (cycle 1st is 28 days, the other cycles are 21 days)
Maximum Concentration (Cmax) of BA1106 | up to cycle 6nd (cycle 1st is 28 days, the other cycles are 21 days)
Minimum Concentration (Cmin) of BA1106 | up to cycle 6nd (cycle 1st is 28 days, the other cycles are 21 days)
Time of maximum concentration (Tmax) of BA1106 | up to cycle 6nd (cycle 1st is 28 days, the other cycles are 21 days)
Clearance (CL) of BA1106 | up to cycle 6nd (cycle 1st is 28 days, the other cycles are 21 days)
Volume of distribution at steady-state conditions (Vss) of BA1106 | up to cycle 6nd (cycle 1st is 28 days, the other cycles are 21 days)
Incidence and titer of Anti-Drug Antibodies (ADA) during the study relative to the prevalence of ADA at baseline | up to 2 years
Incidence of Neutralizing Antibodies (Nab) during the study relative to the prevalence of Nab at baseline | up to 2 years
Objective Response Rate (ORR) | up to 2 years
Duration of Response (DOR) | up to 2 years
Disease Control Rate (DCR) | up to 2 years
Progression-Free Survival (PFS) | up to 2 years
Overall Survival (OS) | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No